CLINICAL TRIAL: NCT01531868
Title: A Randomized Trial of Alternative Sensory Presentation Formats in Asymptomatic Carotid Stenosis
Brief Title: Alternative Sensory Presentation Formats in Asymptomatic Carotid Stenosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Brian Silver, Director, Stroke Center, Rhode Island Hospital
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: ASPFACS-1
Record Dates: First submitted 2012-02-06; First posted 2012-02-13 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Carotid Stenosis
Keywords: Decision making; Carotid stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Auditory qualitative (Other)
  Interventions: Other: Video
- Auditory absolute risk (Other)
  Interventions: Other: Video
- Auditory relative risk (Other)
  Interventions: Other: Video
- Visual qualitative (Other)
  Interventions: Other: Video
- Visual relative risk (Other)
  Interventions: Other: Video
- Visual absolute risk (Other)
  Interventions: Other: Video

INTERVENTIONS:
Other: Video — Video of physician
  Arms: Auditory qualitative
Other: Video — Video of physician
  Arms: Auditory absolute risk
Other: Video — Video of physician
  Arms: Auditory relative risk
Other: Video — Video of physician
  Arms: Visual qualitative
Other: Video — Video of physician
  Arms: Visual relative risk
Other: Video — Video of physician
  Arms: Visual absolute risk

SUMMARY:
Background: In a previous study, information verbally presented as relative risk (e.g. "50% less likely") or qualitative risk (e.g. "significantly less likely") resulted in many more people (66%) choosing a surgical procedure for narrowing or artery in the neck than people presented with absolute risk (e.g. "11% versus 5% over 5 years"), annualized risk (e.g. "2% versus 1% per year for 5 years") and event-free survival (e.g. "95% versus 89% over 5 years") (33%).

Objectives: The purpose of this study is to determine whether the same observations are true for information that is presented visually as a bar graph. In addition, the investigators also seek to determine whether subjects feel that they understand the information better when presented visually as compared with verbally.

Methods: 450 subjects will be approached in the neurology clinic as they are waiting for their office visit. If the subject agrees to participate in this 10 minute study, they will be taken to a quiet room where they will watch a 1 minute video on a laptop. The video will feature an acting physician. The presenter will be the same for all experiment groups. The presenter will describe a hypothetical medical situation in which a narrowing of one of the carotid (neck) arteries is present. The presenter will then describe the risk of a stroke related to that condition if the subject chooses medical therapy versus medical and surgical therapy. The presentation of risk will vary and may be presented in one of 3 different ways including a qualitative description, an absolute risk reduction over a fixed time period, and a relative risk reduction. These three risk groups will be presented either verbally or visually through bar graphs. In the visual subject groups, the presenter will be holding up a graph and remain silent while the graph is shown. The amount of time allotted for the graph on the video will be equal to the amount of time it takes the presenter to say the information in the auditory subject groups. Given that there will be 2 sensory modalities (verbal of visual) and 3 different presentation formats, there will be a total of 6 different videos. After the video is complete, the subject will be asked to complete a 1 page survey which will ask about the patient's age, gender, educational level, reason for the medical visit, and final decision about choice of treatment. The subjects will also answer how well they understood the data by making a mark on a 10 cm horizontal line.

DETAILED DESCRIPTION:
Background: A previous randomized study found that verbal presentation of benefit of surgery in asymptomatic carotid stenosis expressed as qualitative or relative risk resulted in a higher proportion (66% versus 33%) of subjects choosing surgery as compared to subjects presented absolute risk, yearly risk, or event-free survival. Other variables that increased the choice of surgery were male gender, younger age, and higher level of education. Nevertheless, presentation format was the strongest predictor of treatment choice.

Objective/Hypothesis: To determine whether presentation format affects visual representation of information. The investigators hypothesis is that visual representation of both positive and negative outcomes in a single bar graph will result in less subjects favoring surgery as compared to those only shown relative information in a bar graph. The investigators also hypothesize that subjects shown visual information will express a greater understanding of information presented to them as compared to those given verbal information.

Specific Aims: 1) To determine whether presentation format affects visual representation of information. 2) To determine whether subjects given visual representations of information express a greater understanding of the information as compared with subjects given verbal representations of information.

Study Design: 450 subjects will be approached in the neurology clinic as they are waiting for their office visit. Subjects without carotid stenosis will be approached randomly by the principal investigator or one of the co-investigators. They will be asked to participate in the study after completing their office visit with their physician. In the event that the patient is expecting longer than a 30 minute delay to see their physician, they will be asked to participate in the study prior to the office visit. If the subject agrees to participate in this 10 minute study, they will be taken to a quiet room where they will watch a 1 minute video on a laptop. The video will feature an acting physician. The presenter will be the same for all experiment groups. The presenter will describe a hypothetical medical situation in which a narrowing of one of the carotid arteries is present. The presenter will then describe the risk of a stroke related to that condition if the subject chooses medical therapy versus medical and surgical therapy. The presentation of risk will vary and may be presented in one of 3 different ways including a qualitative description, an absolute risk reduction over a fixed time period, and a relative risk reduction. These three risk groups will be presented either verbally or visually through bar graphs. In the visual subject groups, the presenter will be holding up a graph and remain silent while the graph is shown. The amount of time allotted for the graph on the video will be equal to the amount of time it takes the presenter to say the information in the auditory subject groups. Given that there will be 2 sensory modalities (verbal of visual) and 3 different presentation formats, there will be a total of 6 different videos. Randomization will be performed by selecting a video number from an opaque envelope. The subject will be allowed to watch the video up to 3 times, if requested. After the video is complete, the subject will be asked to complete a 1 page survey which will ask about the patient's age, gender, educational level, reason for the medical visit, and final decision about choice of treatment. The subjects will also answer how well they understood the data by making a mark on a 10 cm horizontal line. A mark further to the right signifies better understanding than a mark placed to the left. Data will be entered into a spreadsheet which will then be used to analyze aggregate data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater

Exclusion Criteria:

* No history or carotid stenosis
* No history of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Decision to have surgery | 6 months
  Subjects will complete a survey immediately after watching the video. The completed surveys will then be analyzed after enrollment is complete.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Silver, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Silver B, Zaman IF, Ashraf K, Majed Y, Norwood EM, Schuh LA, Smith BJ, Smith RE, Schultz LR. A randomized trial of decision-making in asymptomatic carotid stenosis. Neurology. 2012 Jan 31;78(5):315-21. doi: 10.1212/WNL.0b013e31824528df. Epub 2012 Jan 4. PMID 22218277